CLINICAL TRIAL: NCT06249373
Title: A Multicenter Randomized Controlled Trial on the Effect of Low-intensity Pulsed Ultrasound on the Maturation of Newly Constructed Autogenous Arteriovenous Fistulas in Uremic Patients
Brief Title: The Effect of LIPUS on the Maturation of Newly Constructed Autogenous AVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Municipal Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Second Affiliated Hospital of Soochow University (Other); Dushu Lake Hospital Affiliated to Soochow University (Other)
Responsible Party: Principal Investigator, Qiang Chen, Head of Nephrology, Suzhou Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-2023-094
Record Dates: First submitted 2024-01-29; First posted 2024-02-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Uremia; Chronic
MeSH Terms: conditions — Uremia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIPUS intervention group (Experimental): Low intensity pulse ultrasound （LIPUS） intervenes at the anastomotic site, and if the ultrasound examination indicates the presence of a narrow site in the outflow tract, it also intervenes at the narrow site. It belongs to non-invasive extracorporeal intervention, with three times a week （during dialysis） for 20 minutes each time. The sound intensity is 350mW/cm2, the pulse frequency is 1MHz, the pulse repetition frequency is 100Hz, the pulse frequency is 100 times, and the treatment period is 12 weeks.
  Interventions: Device: Low intensity pulse ultrasound （LIPUS） intervention for arteriovenous fistula anastomosis
- Simulated LIPUS control group (No Intervention): Using the same forearm wearable portable ultrasound as the LIPUS arteriovenous fistula intervention group, but not issuing low-intensity pulse ultrasound.

INTERVENTIONS:
Device: Low intensity pulse ultrasound （LIPUS） intervention for arteriovenous fistula anastomosis — The LIPUS intervention group for arteriovenous fistula should receive forearm wearable portable low-intensity pulse ultrasound （LIPUS） intervention at the anastomotic site no more than 3 days after suture removal two weeks after the fistula surgery. If the ultrasound examination indicates the presence of stenosis in the outflow tract, the intervention should also be performed at the same time. It belongs to non-invasive extracorporeal intervention, with three times a week （during dialysis） for 20 minutes each time. The sound intensity is 350mW/cm2, the pulse frequency is 1MHz, the pulse repetition frequency is 100Hz, the pulse frequency is 100 times, and the treatment period is 12 weeks.
  Arms: LIPUS intervention group

SUMMARY:
This study aims to evaluate the effect of 12 week low-intensity pulse ultrasound (LIPUS) intervention on the maturation of newly constructed autologous arteriovenous fistulas in uremic patients. This study is a prospective, blinded, randomized controlled trial. This trial is divided into two stages. The first stage is a concept validation trial, which is a single center, prospective, blinded, randomized controlled clinical study. Subjects who meet the screening criteria are randomly divided into an intervention group and a control group in a 1:1 ratio. All subjects underwent safety and efficacy evaluations at the 2nd, 4th, 8th, 12th, and 4th week after treatment. After completing a 4-week follow-up of the 20th study subject, an analysis was conducted with the preset goal of achieving a higher maturation rate of arteriovenous fistula in the intervention group compared to the control group at the follow-up point, and the safety of the study was evaluated. The second stage is a key trial, which is a multicenter, prospective, blinded, randomized controlled clinical study. The inclusion criteria, primary and secondary endpoints, and safety endpoints of the study subjects remain unchanged, and the safety and efficacy of the overall population are evaluated.

ELIGIBILITY:
Inclusion Criteria:

1.18 years old ≤ Age ≤ 75 years old, regardless of gender or ethnicity;

2.Dialysis or non-dialysis patients who have newly established autologous arteriovenous fistula in the wrist and have not yet used the fistula for hemodialysis treatment;

3.Before establishing an autologous arteriovenous fistula in the wrist, ultrasound examination will be performed. The radial artery diameter at the intended surgical site is>1.5mm, and the head vein diameter is>2mm （using a tourniquet）. The arterial and venous blood flow are unobstructed, and the distance between the vein and the skin is<6mm;

4. After introducing dialysis, the calcium ion concentration in the dialysate will be maintained at 1.5mmol/L during the dialysis period, and low molecular weight heparin will be used for anticoagulation. The dosage of low molecular weight heparin remains unchanged （±1000U） during the study period;

5. Sign an informed consent form.

Exclusion Criteria:

1. Poor healing of internal fistula surgical incision;
2. Active bacterial or viral infections;
3. Pregnant women;
4. The patient underwent kidney transplantation or was transferred to peritoneal dialysis during the study period;
5. Subject ALT, AST ≥ 3 × upper limit of normal values;
6. Within 3 months, according to NYHA classification, heart function is classified as level III-IV;
7. Newly diagnosed unstable angina and cerebrovascular events within 3 months;
8. Blood pressure below 90/60mmHg or above 180/100mmHg in the past 2 weeks;
9. During the study period, patients did not follow medical advice and arbitrarily changed the types and dosages of other anticoagulants or anticoagulants (such as aspirin, clopidogrel, Agat Roban, etc.);
10. Combine the use of glucocorticoids and immunosuppressants, such as tacrolimus, cyclosporine, MMF, azathioprine, leflunomide, Tripterygium wilfordii glycosides, etc;
11. Other researchers consider inappropriate situations, such as coexisting with malignant tumors, where the expected lifespan is less than 6 months;
12. I have participated in other clinical trials within 4 weeks prior to the start of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maturity rate of arteriovenous fistula | 12 weeks after enrollment
  Puncture segment venous diameter
Maturity rate of arteriovenous fistula | 12 weeks after enrollment
  Brachial artery blood flow rate

SECONDARY OUTCOMES:
Changes in hemodynamic parameters | 2 weeks,4weeks,8weeks,12weeks after enrollment, and 4 weeks after follow-up.
  Blood flow
Changes in hemodynamic parameters | 2 weeks,4weeks,8weeks,12weeks after enrollment, and 4 weeks after follow-up.
  Minimum outflow venous diameter
Changes in hemodynamic parameters | 2 weeks,4weeks,8weeks,12weeks after enrollment, and 4 weeks after follow-up.
  Primary patency rate
Changes in hemodynamic parameters | 2 weeks,4weeks,8weeks,12weeks after enrollment, and 4 weeks after follow-up.
  Secondary patency rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqing Kong, Study Chair — Suzhou Municipal Hospital; Huijuan Mao, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The Affiliated Suzhou Hospital of Nanjing Medical University, Suzhou Municipal Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunes NS, Chandran P, Sundby M, Visioli F, da Costa Goncalves F, Burks SR, Paz AH, Frank JA. Therapeutic ultrasound attenuates DSS-induced colitis through the cholinergic anti-inflammatory pathway. EBioMedicine. 2019 Jul;45:495-510. doi: 10.1016/j.ebiom.2019.06.033. Epub 2019 Jun 26. PMID 31253515
- [Background] Salmela B, Hartman J, Peltonen S, Alback A, Lassila R. Thrombophilia and arteriovenous fistula survival in ESRD. Clin J Am Soc Nephrol. 2013 Jun;8(6):962-8. doi: 10.2215/CJN.03860412. Epub 2013 Feb 14. PMID 23411429
- [Background] Sifuentes-Franco S, Padilla-Tejeda DE, Carrillo-Ibarra S, Miranda-Diaz AG. Oxidative Stress, Apoptosis, and Mitochondrial Function in Diabetic Nephropathy. Int J Endocrinol. 2018 Apr 1;2018:1875870. doi: 10.1155/2018/1875870. eCollection 2018. PMID 29808088
- [Background] Masengu A, McDaid J, Maxwell AP, Hanko JB. Preoperative radial artery volume flow is predictive of arteriovenous fistula outcomes. J Vasc Surg. 2016 Feb;63(2):429-35. doi: 10.1016/j.jvs.2015.08.106. PMID 26804217
- [Background] Riella MC, Roy-Chaudhury P. Vascular access in haemodialysis: strengthening the Achilles' heel. Nat Rev Nephrol. 2013 Jun;9(6):348-57. doi: 10.1038/nrneph.2013.76. Epub 2013 Apr 16. PMID 23591442
- [Background] Al-Jaishi AA, Oliver MJ, Thomas SM, Lok CE, Zhang JC, Garg AX, Kosa SD, Quinn RR, Moist LM. Patency rates of the arteriovenous fistula for hemodialysis: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Mar;63(3):464-78. doi: 10.1053/j.ajkd.2013.08.023. Epub 2013 Oct 30. PMID 24183112
- [Background] Dember LM, Beck GJ, Allon M, Delmez JA, Dixon BS, Greenberg A, Himmelfarb J, Vazquez MA, Gassman JJ, Greene T, Radeva MK, Braden GL, Ikizler TA, Rocco MV, Davidson IJ, Kaufman JS, Meyers CM, Kusek JW, Feldman HI; Dialysis Access Consortium Study Group. Effect of clopidogrel on early failure of arteriovenous fistulas for hemodialysis: a randomized controlled trial. JAMA. 2008 May 14;299(18):2164-71. doi: 10.1001/jama.299.18.2164. PMID 18477783
- [Background] Irish AB, Viecelli AK, Hawley CM, Hooi LS, Pascoe EM, Paul-Brent PA, Badve SV, Mori TA, Cass A, Kerr PG, Voss D, Ong LM, Polkinghorne KR; Omega-3 Fatty Acids (Fish Oils) and Aspirin in Vascular Access Outcomes in Renal Disease (FAVOURED) Study Collaborative Group. Effect of Fish Oil Supplementation and Aspirin Use on Arteriovenous Fistula Failure in Patients Requiring Hemodialysis: A Randomized Clinical Trial. JAMA Intern Med. 2017 Feb 1;177(2):184-193. doi: 10.1001/jamainternmed.2016.8029. PMID 28055065
- [Background] Remuzzi A, Bozzetto M, Brambilla P. Is shear stress the key factor for AVF maturation? J Vasc Access. 2017 Mar 6;18(Suppl. 1):10-14. doi: 10.5301/jva.5000686. Epub 2017 Mar 5. PMID 28297046
- [Background] Dolan JM, Kolega J, Meng H. High wall shear stress and spatial gradients in vascular pathology: a review. Ann Biomed Eng. 2013 Jul;41(7):1411-27. doi: 10.1007/s10439-012-0695-0. Epub 2012 Dec 11. PMID 23229281
- [Background] Kaygin MA, Halici U, Aydin A, Dag O, Binici DN, Limandal HK, Arslan U, Kiymaz A, Kahraman N, Calik ES, Savur AI, Erkut B. The relationship between arteriovenous fistula success and inflammation. Ren Fail. 2013 Sep;35(8):1085-8. doi: 10.3109/0886022X.2013.815100. Epub 2013 Aug 1. PMID 23906289
- [Background] Asare Y, Schmitt M, Bernhagen J. The vascular biology of macrophage migration inhibitory factor (MIF). Expression and effects in inflammation, atherogenesis and angiogenesis. Thromb Haemost. 2013 Mar;109(3):391-8. doi: 10.1160/TH12-11-0831. Epub 2013 Jan 17. PMID 23329140
- [Background] Stangenberg S, Nguyen LT, Chen H, Al-Odat I, Killingsworth MC, Gosnell ME, Anwer AG, Goldys EM, Pollock CA, Saad S. Oxidative stress, mitochondrial perturbations and fetal programming of renal disease induced by maternal smoking. Int J Biochem Cell Biol. 2015 Jul;64:81-90. doi: 10.1016/j.biocel.2015.03.017. Epub 2015 Apr 4. PMID 25849459
- [Background] Yang B, Janardhanan R, Vohra P, Greene EL, Bhattacharya S, Withers S, Roy B, Nieves Torres EC, Mandrekar J, Leof EB, Mukhopadhyay D, Misra S. Adventitial transduction of lentivirus-shRNA-VEGF-A in arteriovenous fistula reduces venous stenosis formation. Kidney Int. 2014 Feb;85(2):289-306. doi: 10.1038/ki.2013.290. Epub 2013 Aug 7. PMID 23924957
- [Background] Veillat V, Carli C, Metz CN, Al-Abed Y, Naccache PH, Akoum A. Macrophage migration inhibitory factor elicits an angiogenic phenotype in human ectopic endometrial cells and triggers the production of major angiogenic factors via CD44, CD74, and MAPK signaling pathways. J Clin Endocrinol Metab. 2010 Dec;95(12):E403-12. doi: 10.1210/jc.2010-0417. Epub 2010 Sep 8. PMID 20829186
- [Background] Stracke S, Konner K, Kostlin I, Friedl R, Jehle PM, Hombach V, Keller F, Waltenberger J. Increased expression of TGF-beta1 and IGF-I in inflammatory stenotic lesions of hemodialysis fistulas. Kidney Int. 2002 Mar;61(3):1011-9. doi: 10.1046/j.1523-1755.2002.00191.x. PMID 11849456
- [Background] Dukkipati R, Molnar MZ, Park J, Jing J, Kovesdy CP, Kajani R, Kalantar-Zadeh K. Association of vascular access type with inflammatory marker levels in maintenance hemodialysis patients. Semin Dial. 2014 Jul-Aug;27(4):415-23. doi: 10.1111/sdi.12146. Epub 2013 Oct 9. PMID 24118625
- [Background] Vassalotti JA, Jennings WC, Beathard GA, Neumann M, Caponi S, Fox CH, Spergel LM; Fistula First Breakthrough Initiative Community Education Committee. Fistula first breakthrough initiative: targeting catheter last in fistula first. Semin Dial. 2012 May;25(3):303-10. doi: 10.1111/j.1525-139X.2012.01069.x. Epub 2012 Apr 4. PMID 22487024
- [Background] Lin CC, Chang CF, Lai MY, Chen TW, Lee PC, Yang WC. Far-infrared therapy: a novel treatment to improve access blood flow and unassisted patency of arteriovenous fistula in hemodialysis patients. J Am Soc Nephrol. 2007 Mar;18(3):985-92. doi: 10.1681/ASN.2006050534. Epub 2007 Jan 31. PMID 17267744
- [Background] Gigliotti JC, Huang L, Ye H, Bajwa A, Chattrabhuti K, Lee S, Klibanov AL, Kalantari K, Rosin DL, Okusa MD. Ultrasound prevents renal ischemia-reperfusion injury by stimulating the splenic cholinergic anti-inflammatory pathway. J Am Soc Nephrol. 2013 Sep;24(9):1451-60. doi: 10.1681/ASN.2013010084. Epub 2013 Aug 1. PMID 23907510
- [Background] Charles EJ, Tian Y, Zhang A, Wu D, Mehaffey JH, Gigliotti JC, Klibanov AL, Kron IL, Yang Z. Pulsed ultrasound attenuates the hyperglycemic exacerbation of myocardial ischemia-reperfusion injury. J Thorac Cardiovasc Surg. 2021 Apr;161(4):e297-e306. doi: 10.1016/j.jtcvs.2019.10.096. Epub 2019 Nov 2. PMID 31839230
- [Background] Zachs DP, Offutt SJ, Graham RS, Kim Y, Mueller J, Auger JL, Schuldt NJ, Kaiser CRW, Heiller AP, Dutta R, Guo H, Alford JK, Binstadt BA, Lim HH. Noninvasive ultrasound stimulation of the spleen to treat inflammatory arthritis. Nat Commun. 2019 Mar 12;10(1):951. doi: 10.1038/s41467-019-08721-0. PMID 30862842
- [Background] Xu T, Gu J, Li C, Guo X, Tu J, Zhang D, Sun W, Kong X. Low-intensity pulsed ultrasound suppresses proliferation and promotes apoptosis via p38 MAPK signaling in rat visceral preadipocytes. Am J Transl Res. 2018 Mar 15;10(3):948-956. eCollection 2018. PMID 29636884
- [Background] Su Z, Xu T, Wang Y, Guo X, Tu J, Zhang D, Kong X, Sheng Y, Sun W. Low-intensity pulsed ultrasound promotes apoptosis and inhibits angiogenesis via p38 signaling-mediated endoplasmic reticulum stress in human endothelial cells. Mol Med Rep. 2019 Jun;19(6):4645-4654. doi: 10.3892/mmr.2019.10136. Epub 2019 Apr 5. PMID 30957188
- [Background] Toyama Y, Sasaki K, Tachibana K, Ueno T, Kajimoto H, Yokoyama S, Ohtsuka M, Koiwaya H, Nakayoshi T, Mitsutake Y, Chibana H, Itaya N, Imaizumi T. Ultrasound stimulation restores impaired neovascularization-related capacities of human circulating angiogenic cells. Cardiovasc Res. 2012 Sep 1;95(4):448-59. doi: 10.1093/cvr/cvs173. Epub 2012 May 28. PMID 22641844